CLINICAL TRIAL: NCT03070678
Title: Open-label, Cross Over, Single-sequence, Two Periods Phase 1 Drug-drug Interaction Study to Evaluate the Effects of Multiple-dose Mefenamic Acid, a Known UGT1A9 Inhibitor, on the Pharmacokinetics and Pharmacodynamics of Single-dose Sotagliflozin in Healthy Male and Female Subjects
Brief Title: Interaction Study to Evaluate the Effects of Mefenamic Acid on the Pharmacokinetics and Pharmacodynamics of Sotagliflozin in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INT14937; U1111-1186-2702 (Other: UTN)
Record Dates: First submitted 2017-02-21; First posted 2017-03-03 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Mefenamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR439954 with or without mefenamic acid (Experimental): Period 1: single oral dose of 400 mg sotagliflozin Period 2: initial loading dose of 500 mg in the morning of Day 1, followed by 250 mg from Day 1 H6 to Day 7 of mefenamic acid and a single oral dose of sotagliflozin on Day 2
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Mefenamic acid

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Mefenamic acid — Pharmaceutical form: capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the effect of multiple dose mefenamic acid on the pharmacokinetics (PK) of sotagliflozin and its metabolite in healthy male and female subjects.

Secondary Objectives:

* To assess total 24 hour urinary glucose excretion (UGE) after 400 mg sotagliflozin alone and in combination with mefenamic acid in healthy male and female subjects.
* To assess the safety and tolerability of sotagliflozin alone and in combination with mefenamic acid in healthy male and female subjects.

DETAILED DESCRIPTION:
The expected duration of the study is approximately 59 days per subject, including 2-28 days of screening, treatment period 1 of 7 days, treatment period 2 of 8 days, at least 7 days of wash-out period, and an end of study visit, which is between 14-21 days after the last dose of sotagliflozin.

ELIGIBILITY:
Inclusion criteria :

* Healthy male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, ECG, and laboratory parameters, aPTT (activated partial thromboplastin time) should not exceed normal control more than 10 seconds.
* Female subject must use a double contraception method including a highly effective method of birth control except if she has undergone sterilization at least 3 months earlier or is postmenopausal.
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.

Exclusion criteria:

* Any history or presence of clinically relevant disease at screening, which could interfere with the objectives of the study or the safety of the subject's participation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive β-HCG (human chorionic gonadotropin) blood test if applicable), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion. Any oral contraceptives during the screening period or for at least 15 days prior to inclusion; any injectable contraceptives or hormonal intrauterine devices within 12 months prior to inclusion; or topical controlled delivery contraceptives (patch) for 3 months prior to inclusion.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 144 hours after each SAR439954 intake
Area under the concentration-time curve from 0 to the last quantifiable concentration (AUClast) | Up to 144 hours after each SAR439954 intake
Area under the concentration-time curve from 0 to infinity (AUC0 ∞) | Up to 144 hours after each SAR439954 intake

SECONDARY OUTCOMES:
Total 24-hour UGE (urinary glucose excretion) after each dose with sotagliflozin | Up to 24 hours after each SAR439954 intake

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site 250001, Gières, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org